CLINICAL TRIAL: NCT00997906
Title: A Randomised Phase II/III Study of Concurrent Cisplatin-Radiotherapy With or Without Induction Chemotherapy Using Gemcitabine, Carboplatin and Paclitaxel in Locally Advanced Nasopharyngeal Cancer
Brief Title: Cisplatin and RT With or Without Gemcitabine, Carboplatin, and Paclitaxel in Treating Patients With Locally Advanced NPC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Principal Investigator, Terence Tan Wee Kiat, Senior Consultant, National Cancer Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000657121; SINGAPORE-NCC0901 (Other: National Cancer Centre Singapore)
Record Dates: First submitted 2009-10-17; First posted 2009-10-20 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Head and Neck Cancer
Keywords: stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Carboplatin; Cisplatin; Gemcitabine; Paclitaxel; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive cisplatin IV over 2 hours once weekly on weeks 1-8 and undergo intensity-modulated radiotherapy once daily, 5 days a week, on weeks 1-7 (6½ weeks for a total of 33 fractions).
  Interventions: Drug: cisplatin; Radiation: intensity-modulated radiation therapy
- Arm II (Experimental): Patients receive induction chemotherapy comprising gemcitabine hydrochloride IV over 30 minutes, carboplatin IV over 1 hour, and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 3 courses. Beginning at least 3 weeks after the last dose of induction chemotherapy, patients receive cisplatin and undergo radiotherapy as in arm I.
  Interventions: Drug: carboplatin,; Drug: cisplatin; Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Drug: carboplatin, — Given IV
  Arms: Arm II
Drug: cisplatin — Given IV
Drug: gemcitabine hydrochloride — Given IV
  Arms: Arm II
Drug: paclitaxel — Given IV
  Arms: Arm II
Radiation: intensity-modulated radiation therapy — Given once daily 5 days a week for 6½ weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, gemcitabine hydrochloride, carboplatin, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy together with radiation therapy my kill more tumor cells. It is not yet known whether giving cisplatin together with radiation therapy is more effective with or without gemcitabine hydrochloride, carboplatin, and paclitaxel in treating patients with nasopharyngeal cancer.

PURPOSE: This randomized phase II/III trial is studying how well giving cisplatin together with radiation therapy works compared with giving cisplatin and radiation therapy together with gemcitabine hydrochloride, carboplatin, and paclitaxel in treating patients with locally advanced nasopharyngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the 5-year overall survival of patients with locally advanced nasopharyngeal cancer treated with concurrent cisplatin and radiotherapy with vs without induction chemotherapy comprising gemcitabine hydrochloride, carboplatin, and paclitaxel.

Secondary

* To assess and compare the disease-free survival, distant metastases rate, toxicities, and quality of life of patients treated with these regimens.

OUTLINE: Patients are stratified by N-stage (N0-1 vs N2-3) and are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cisplatin IV over 2 hours once weekly on weeks 1-8 and undergo intensity-modulated radiotherapy once daily, 5 days a week, on weeks 1-7 (6½ weeks for a total of 33 fractions).
* Arm II: Patients receive induction chemotherapy comprising gemcitabine hydrochloride IV over 30 minutes, carboplatin IV over 1 hour, and paclitaxel IV over 1 hour on days 1 and 8. Treatment repeats every 21 days for 3 courses. Beginning at least 3 weeks after the last dose of induction chemotherapy, patients receive cisplatin and undergo radiotherapy as in arm I.

Quality of life is assessed periodically.

After completion of study treatment, patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion criteria:

Patients are eligible for inclusion if all of the following criteria are fulfilled:

1. Have given written informed consent, with the understanding that consent may be withdrawn at any time without prejudice.
2. Loco-regional advanced NPC UICC (1997) Stages T3 - 4 any N, or any Stage T, N2 - 3.
3. A histological diagnosis of WHO Type II or III NPC must have been established at some time and the investigator must review and confirm the diagnosis prior to randomization.
4. No evidence of distant metastases in staging work up (including lung, liver and bone imaging).
5. Cross sectional imaging of the primary and neck disease (MRI preferred)
6. Evaluable disease must be present.
7. Performance status of ECOG grade 0 or 1 (see Appendix I).
8. No prior tumour therapy
9. Adequate bone marrow, renal and hepatic function:

   Bone marrow : WBC > 3000 / mm3 (ANC > 1500 / mm3 ),
   * Platelets > 100 000 / mm3,
   * Hb > 10 gm/dl Renal : serum creatinine within institutional normal range (or) lower than the lower limit of institutional normal range
   * calculated creatinine clearance > 50 ml / min Hepatic : enzymes (SAP, SGOT) < 2x normal
   * bilirubin < 24 µmol / l.
10. At least 18 years of age, of either sex.

Exclusion criteria:

Patients are to be excluded from the study if any of the following criteria is fulfilled:

1. Uncontrolled hypercalcaemia: calcium ≥ 2.7 mmol/L (10.8 mg/dL).
2. Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin).
3. Other serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
4. Have serious active infection.
5. Hepatitis B carrier
6. Prior treatment including chemotherapy or radiotherapy.
7. Pregnant or lactating female subjects and subjects with reproductive potential not implementing adequate contraceptive measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2009-09-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 5 years | 5 years

SECONDARY OUTCOMES:
Metastases-free survival | 10 years
Disease-free survival | 10 years
Tumor recurrence | 10 years
Toxicity according to the Common Toxicity Criteria | 10 years
Quality of life as measured by the EORTC QLQ-C30 | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Terence Tan, FRCR, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No